CLINICAL TRIAL: NCT05612126
Title: Pre- and Post-tests Impact of a Football Tournament on the Mental Well-being of Kuru Community Youths in Jos-South: A Single Arm Mixed Methods Study
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Nottingham Trent University (Other)
Collaborators: Teesside University (Other); Coal City University (Unknown); Dung Jidong Foundation (Unknown)
Responsible Party: Principal Investigator, Dr Dung Jidong, PhD, Senior Lecturer, Nottingham Trent University
Other Study IDs: 0000-0001-5034-0335c
Record Dates: First submitted 2022-11-03; First posted 2022-11-10 (Actual); Last update posted 2022-11-10 (Actual); Status verified 2022-11

CONDITIONS: Football Tournament

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Sporting activities such as football tournaments are instrumental in promoting community mental health. A community-based football tournament intervention will benefit the participating individuals' physical and mental health and promote community cohesion.

The anticipated benefits of the proposed football tournament are:

* To bring a greater sense of community cohesion and togetherness.
* To improve physical and mental health (e.g., increase fitness, reduce anxiety, depression, loneliness, suicidal ideation or self-harm).

ELIGIBILITY:
Inclusion Criteria:

* Male youths
* Between 18 and 35 years
* Able to give informed consent
* Residents of the Kuru community of Jos-South
* No history of chronic health concerns (e.g., chronic heart disease, severe depression etc).

Exclusion Criteria:

* Females
* Below 18 or above 35 years
* Unable to give informed consent
* History of chronic health concerns (e.g., chronic heart disease, severe depression etc).

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Male youths football tournament intervention
Study Population: Kuru community male youths in Jos-South local government area of Plateau State Nigeria.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2022-11-21 (Estimated); Primary Completion 2023-11-20 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in Football Worry is being assessed | Change is being assessed at pre and post-intervention at 8 weeks
  Primary outcome measure would be assessed using the Football Worry Scale
Change in Moral Disengagement in Sport is being assessed | Change is being assessed at pre and post-intervention at 8 weeks
  Primary outcome measure would be assessed using the Moral Disengagement in Sport Scale
Change in Positive Mental Health is being assessed | Change is being assessed at pre and post-intervention at 8 weeks
  Primary outcome measure would be assessed using the Positive Mental Health Scale
Change in Psychological Well-Being is being assessed | Change is being assessed at pre and post-intervention at 8 weeks
  Primary outcome measure would be assessed using the Psychological Well-Being Measure

IPD SHARING:
Plan to Share IPD: Yes